CLINICAL TRIAL: NCT03959137
Title: BEPACT Lung: Impact of Patient Characteristics on Pneumo-oncologists Non Small Cell Lung Cancer (NSCLC) Systemic Treatment Decision in Belgium: A Cross-sectional Study
Brief Title: BEPACT- Lung: Impact of Patient Characteristics on Pneumo-oncologists Non Small Cell Lung Cancer (NSCLC) Systemic Treatment Decision in Belgium
Acronym: BEPACT- Lung
Status: Completed | Type: Observational
Sponsor: MSD Belgium BVBA (Industry)
Responsible Party: Sponsor
Other Study IDs: VEAP7678
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-03

CONDITIONS: Stage IV Non-small Cell Lung Cancer
Keywords: Treatment choice
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary study group: Stage IV untreated NSCLC
  Interventions: Other: None - Common practice

INTERVENTIONS:
Other: None - Common practice — None - Common practice

SUMMARY:
The treatment landscape of metastatic non small cell lung cancer (NSCLC) is rapidly evolving. There are new diagnostic and treatment options available in the coming months and years.

New combination treatments will give different solutions to pneumo-oncologists who might be guided by certain patient and tumor characteristics.

The link between patient and tumor characteristics in untreated stage IV non small cell lung cancer (NSCLC) patients and systemic treatment needs further investigation, allowing the identification of possible treatment issues, data gaps and/or areas of improvement.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional, cross-sectional study. Consecutive patients with metastatic stage IV non small cell lung cancer (NSCLC) selected for systemic treatment or best supportive care will be included in the trial at the time the patient signed the informed consent form (ICF). Patients that were selected for systemic treatment, should have received at least their first dose and a maximum of one cycle of the same treatment.

The pneumo-oncologist that treats the patient will fill in the CRF, indicating the systemic treatment option and the link with the variable categories that impacted the choice for a systemic treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Have voluntarily agreed to participate by giving written informed consent/assent for the trial.
* Have a histologically or cytologically confirmed diagnosis of stage IV non-small cell lung cancer (NSCLC) on first-line (1L) systemic treatment.
* Have received at least their first dose of the selected systemic treatment and a maximum of 1 cycle of the same treatment. Patients that were selected to receive best supportive care will not have to comply to this inclusion criterion.
* Be ≥ 18 years of age on day of signing informed consent.

Exclusion Criteria:

* Has received prior systemic treatment for their metastatic non-small cell lung cancer (NSCLC) before the first dose of trial treatment. However, subjects who received adjuvant or neoadjuvant therapy during an earlier stage of their disease, but evolved to stage IV, are eligible.
* Tyrosine kinase inhibitor (TKI) selected as first-line systemic treatment.
* Is participating in an interventional trial or medical need program.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: At least 200 stage IV non-small cell lung cancer (NSCLC)subjects treated in approximately 20 Belgian hospitals starting first-line treatment or best supportive care will be enrolled in line with inclusion and exclusion criteria. Assuming that three stage IV NSCLC subjects can be recruited per month per site, enrollment period has been set to 5 months. Only a maximum of 10% of subjects can be enrolled by one site.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- Belgium (21):
  - UZA, Antwerp
  - ZNA Middelheim, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - CHIREC, Brussels
  - Cliniques Universitaires Saint-Luc UCL Bruxelles, Brussels
  - UZ Brussel, Brussels
  - CH de Charleroi, Charleroi
  - UZ Gent, Ghent
  - CH Jolimont, Haine-Saint-Paul
  - Jessa Ziekenhuis, Hasselt
  - Az Groeninghe Kortrijk, Kortrijk
  - UZ Leuven, Leuven
  - CHC Liège, Liège
  - CHR Citadelle, Liège
  - CHU de Liège, Liège
  - CHU UCL Namur, site Godinne, Namur
  - Clinique St-Pierre Ottignies, Ottignies
  - AZ Delta, Roeselare
  - AZ St Nikolaas, Saint-Nicolas
  - St Trudo Ziekenhuis, Sint-Truiden
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Study Group - Single Arm: Stage IV untreated non-small cell lung cancer (NSCLC)
  Patient disposition:
  * Enrolled patients n=215
  * Eligible patients n=209
  Total of 215 patients were enrolled in the study at 21 different sites between 03 June 2019 and 31 October 2019.
  Of the enrolled patients, 209 qualified for inclusion in the Eligible Population (i.e. had given informed consent and satisfied all inclusion criteria and none of the exclusion criteria)
Period: Overall Study
Arm/Group | Primary Study Group - Single Arm
Started | 215
Completed | 209
Not Completed | 6
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Groups:
- Primary Study Group: A total of 215 patients were enrolled in the study and 209 qualified for inclusion in the Eligible Population (i.e. had given informed consent and satisfied all inclusion criteria and none of the exclusion criteria).
  All analyses were performed on the Eligible Population.
  * Demography data
  * Age (years)
  * Gender (male or female)
  * Weight loss (%)
  * Smoking status (current, former (defined as smoking ≥ 1 year), never, or unknown)
  * ECOG status (0, 1, 2, 3-4, or unknown)
  * Patient's preference for treatment choice (yes, no, or unknown)
Arm/Group | Primary Study Group
Number analyzed (Participants) | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 136
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Histology [Count of Participants; unit: Participants] — Histology of non small cell lung cancer patients can be divided in squamous, non-squamous, not otherwise specified.
  Participants
    Squamous | 57
    Non-squamous | 137
    Not otherwise specified | 15
ECOG [Count of Participants; unit: Participants] — The ECOG performance status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. Ranging from 0 (fully active) to 5 (dead).
  Participants
    ECOG 0 | 40
    ECOG 1 | 121
    ECOG 2 | 34
    ECOG 3-4 | 11
    Unknown | 3
Smoking Status [Count of Participants; unit: Participants] — Smoking status is definde as current, former (former smoker defined as ≥ 1 year), never, or unknown
  Participants
    Current | 99
    Former (>1 year) | 101
    Never | 8
    Unknown | 1
IHC PD-L1 [Count of Participants; unit: Participants] — Clinical trials have shown the association of programmed cell death 1 (PD-L1) expression by immunohistochemistry (IHC) with higher overall response rates to the PD-1/PD-L1 axis blockade suggesting that PD-L1 expression may serve as a predictive marker.
  Participants
    Tumor Proportion Score (TPS) <1% | 69
    Tumor Proportion Score (TPS) 1-49% | 45
    Tumor Proportion Score (TPS) >=50% | 88
    Unknown | 7

OUTCOME MEASURES:

1. Primary Outcome: The Study Outcome is Defined as the Systemic Treatment Choice.
Description: Systemic treatment choices are defined as :
  1. Chemotherapy (chemo)
  2. Immunotherapy (IO)
  3. immuno combined therapies (IO+IO)
  4. IO+chemo
  5. IO+bevacizumab+chemo (IO+bev+chemo)
  6. best supportive care (BSC). There is no exposure in this study.
Time Frame: during visits 1 and 2, up to approximately 3 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Primary Study Group: Confirmed diagnosis of stage IV NSCLC on first-line (1L) systemic treatment
Arm/Group | Primary Study Group
Number analyzed (Participants) | 209
Participants
  Chemotherpay | 26
  Immunotherapy | 68
  Immunotherapy combined therapies | 0
  Immunotherapy + chemotherapy | 99
  Immunotherapy + bevacizumab + chemotherapy | 0
  Best supportive care | 16

ADVERSE EVENTS:
Time Frame: Timeframe between Visit 1 and 2 varied between same day (0 days in between) and 3 weeks maximum.
Description: Adverse Event Reporting INVESTIGATOR RESPONSIBILITY: If the investigator becomes aware of any serious adverse event (SAE), including death due to any cause, or non-serious adverse reaction (NSAR) following the use of any Merck product, the event must be reported according to Table 1. The investigator must evaluate each SAE for causality and record causality on the AE form for each event reported.
Groups:
- Primary Study Group - Single Arm: This is a primary data collection non-interventional study being conducted within routine medical practice.
  All direction for medication usage is at the discretion of a physician in accordance with usual medical practice.
  No administration of any therapeutic or prophylactic agent is required in this protocol, and there are no procedures required as part of this protocol.
Arm/Group | Primary Study Group - Single Arm
All-Cause Mortality (participants affected / at risk) | 4/215
Serious Adverse Events (participants affected / at risk) | 13/215
Other Adverse Events (participants affected / at risk) | 1/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Study Group - Single Arm (N=215)
Hospitalization (Gastrointestinal disorders) | 3 (3)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 4 (4)
pericardial fluid accumulation (Cardiac disorders) | 1 (1)
Worsened general condition (General disorders) | 2 (2)
Brain metastasis (progression) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Inflammatory folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hospitalisation (General disorders) | 1 (1)
Eosinophelia (Blood and lymphatic system disorders) | 1 (1)
Hospitalization (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Study Group - Single Arm (N=215)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Cutaneous eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Eosinophelia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The experiment is not interventional and cross sectional.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT03959137/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03959137/SAP_001.pdf